CLINICAL TRIAL: NCT02613520
Title: Clinical Trial to Evaluate the Safety and Immunogenicity in Age De-Escalation of Direct Venous Inoculation of a Plasmodium Falciparum Sporozoite Vaccine in Tanzanian Adults, Children, and Infants
Brief Title: Safety and Immunogenicity in Age De-Escalation of PfSPZ Vaccine in Tanzanian Adults, Children, and Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Ifakara Health Institute (Other); Swiss Tropical & Public Health Institute (Other); Medical Care Development, Inc. (Other); Tanzania Commission for Science and Technology (Other); Government of Equatorial Guinea (Other Government); Marathon Oil Corporation (Industry); Noble Oil Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BSPZV2
Record Dates: First submitted 2015-11-17; First posted 2015-11-24 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2017-12

CONDITIONS: Malaria
Keywords: PfSPZ Vaccine; Plasmodium falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (23):
- Group 1a (PfSPZ Vaccine) (Experimental): 18- 45 years; n=6; 3 doses of 9 x 10^5 PfSPZ Vaccine given 8 weeks apart. Volunteers will undergo CHMI with PfSPZ Challenge 3 weeks after the last immunization.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (for CHMI)
- Group 1a (normal saline) (Placebo Comparator): 18- 45 years; n=3; 3 doses of normal saline given 8 weeks apart. Volunteers will undergo CHMI with PfSPZ Challenge 3 weeks after the last immunization.
  Interventions: Other: Normal Saline; Biological: PfSPZ Challenge (for CHMI)
- Group 1a (CHMI controls) (Other): 18- 45 years; n=6; volunteers will not receive any intervention, but will serve only as infectivity controls; 3 volunteers each, for CHMI 1 and for CHMI 2 in Group 1a. Volunteers will be injected with PfSPZ Challenge (for CHMI).
  Interventions: Biological: PfSPZ Challenge (for CHMI)
- Group 1b (PfSPZ Vaccine) (Experimental): 18- 45 years; n=6; 3 doses of 1.8 x 10^6 PfSPZ Vaccine given 8 weeks apart. Volunteers will undergo CHMI with PfSPZ Challenge 3 weeks after the last immunization.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (for CHMI)
- Group 1b (normal saline) (Placebo Comparator): 18- 45 years; n=3; 3 doses of normal saline given 8 weeks apart. Volunteers will undergo CHMI with PfSPZ Challenge 3 weeks after the last immunization.
  Interventions: Other: Normal Saline; Biological: PfSPZ Challenge (for CHMI)
- Group 1b (CHMI controls) (Other): 18- 45 years; n=6; volunteers will not receive any intervention, but will serve only as infectivity controls; 3 volunteers each, for CHMI 1 and for CHMI 2 in Group 1b. Volunteers will be injected with PfSPZ Challenge (for CHMI).
  Interventions: Biological: PfSPZ Challenge (for CHMI)
- Group 2a (PfSPZ Vaccine) (Experimental): 11-17 years; n=6; 3 doses of 9.0 x 10^5 PfSPZ Vaccine given 8 weeks apart.
  Interventions: Biological: PfSPZ Vaccine
- Group 2a (normal saline) (Placebo Comparator): 11-17 years; n=3; 3 doses of normal saline given 8 weeks apart.
  Interventions: Other: Normal Saline
- Group 2b (PfSPZ Vaccine) (Experimental): 11-17 years; n=6; 3 doses of 1.8 x 10^6 PfSPZ Vaccine given 8 weeks apart.
  Interventions: Biological: PfSPZ Vaccine
- Group 2b (normal saline) (Placebo Comparator): 11-17 years; n=3; 3 doses of normal saline given 8 weeks apart.
  Interventions: Other: Normal Saline
- Group 3a (PfSPZ Vaccine) (Experimental): 6-10 years; n=6; 3 doses of 9.0 x 10^5 PfSPZ Vaccine given 8 weeks apart.
  Interventions: Biological: PfSPZ Vaccine
- Group 3a (normal saline) (Placebo Comparator): 6-10 years; n=3; 3 doses of normal saline given 8 weeks apart.
  Interventions: Other: Normal Saline
- Group 3b (PfSPZ Vaccine) (Experimental): 6-10 years; n=6; 3 doses of 1.8 x 10^6 PfSPZ Vaccine given 8 weeks apart.
  Interventions: Biological: PfSPZ Vaccine
- Group 3b (normal saline) (Placebo Comparator): 6-10 years; n=3; 3 doses of normal saline given 8 weeks apart.
  Interventions: Other: Normal Saline
- Group 4a (PfSPZ Vaccine) (Experimental): 1-5 years; n=6; 3 doses of 4.5 x 10^5 PfSPZ Vaccine given 8 weeks apart.
  Interventions: Biological: PfSPZ Vaccine
- Group 4a (normal saline) (Placebo Comparator): 1-5 years; n=3; 3 doses of normal saline given 8 weeks apart.
  Interventions: Other: Normal Saline
- Group 4b (PfSPZ Vaccine) (Experimental): 1-5 years; n=6; 3 doses of 9.0 x 10^5 PfSPZ Vaccine given 8 weeks apart.
  Interventions: Biological: PfSPZ Vaccine
- Group 4b (normal saline) (Placebo Comparator): 1-5 years; n=3; 3 doses of normal saline given 8 weeks apart.
  Interventions: Other: Normal Saline
- Group 5a (PfSPZ Vaccine) (Experimental): 6-11 months; n=3; 1 dose of 2.7 x 10^5 PfSPZ Vaccine.
  Interventions: Biological: PfSPZ Vaccine
- Group 5b (PfSPZ Vaccine) (Experimental): 6-11 months; n=6; 3 doses of 4.5 x 10^5 PfSPZ Vaccine given 8 weeks apart.
  Interventions: Biological: PfSPZ Vaccine
- Group 5b (normal saline) (Placebo Comparator): 6-11 months; n=3; 3 doses of normal saline given 8 weeks apart.
  Interventions: Other: Normal Saline
- Group 5c (PfSPZ Vaccine) (Experimental): 6-11 months; n=6; 3 doses of 9.0 x 10^5 PfSPZ Vaccine given 8 weeks apart.
  Interventions: Biological: PfSPZ Vaccine
- Group 5c (normal saline) (Placebo Comparator): 6-11 months; n=3; 3 doses of normal saline given 8 weeks apart.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: PfSPZ Vaccine — Metabolically active, non-replicating, radiation attenuated, aseptic, purified, cryopreserved NF54 P. falciparum (Pf) sporozoites (PfSPZ Vaccine)
  Arms: Group 1a (PfSPZ Vaccine); Group 1b (PfSPZ Vaccine); Group 2a (PfSPZ Vaccine); Group 2b (PfSPZ Vaccine); Group 3a (PfSPZ Vaccine); Group 3b (PfSPZ Vaccine); Group 4a (PfSPZ Vaccine); Group 4b (PfSPZ Vaccine); Group 5a (PfSPZ Vaccine); Group 5b (PfSPZ Vaccine); Group 5c (PfSPZ Vaccine)
Other: Normal Saline — 0.9% Sodium chloride
  Arms: Group 1a (normal saline); Group 1b (normal saline); Group 2a (normal saline); Group 2b (normal saline); Group 3a (normal saline); Group 3b (normal saline); Group 4a (normal saline); Group 4b (normal saline); Group 5b (normal saline); Group 5c (normal saline)
Biological: PfSPZ Challenge (for CHMI) — live, infectious, aseptic, purified, cryopreserved NF54 P. falciparum (Pf) sporozoites (PfSPZ Challenge) Controlled human malaria infection (CHMI) by direct venous inoculation of 3,200 PfSPZ Challenge
  Arms: Group 1a (CHMI controls); Group 1a (PfSPZ Vaccine); Group 1a (normal saline); Group 1b (CHMI controls); Group 1b (PfSPZ Vaccine); Group 1b (normal saline)

SUMMARY:
The present trial will evaluate safety and tolerability as well as the vaccine-induced humoral and cellular immune responses in healthy Tanzanian adults, adolescents, children, and infants who receive doses of 1.8x10^6, 9.0x10^5, 4.5x10^5 or 2.7x10^5 PfSPZ of PfSPZ Vaccine by direct venous inoculation (DVI),compared with control groups receiving normal saline (NS) placebo by DVI. In addition, as an exploratory objective, controlled human malaria infection (CHMI) will be used to assess efficacy in adults three weeks following immunization.

DETAILED DESCRIPTION:
This is a single center trial to assess the safety, tolerability and immunogenicity of PfSPZ Vaccine administered by direct venous inoculation (DVI) to healthy Tanzanian adults, adolescents, and children and infants. 105 healthy male and female; adults, adolescents, children and infant volunteers, aged from 6 months to 45 years, who live in the Bagamoyo Township will be enrolled based on pre-defined inclusion and exclusion criteria implemented according to international ethical standards.

The safety and tolerability of PfSPZ Vaccine administered as three doses of either 9.0x10^5 PfSPZ or 1.8x10^6 PfSPZ to healthy Tanzanian adults, adolescents, and children 6 years of age or older; and three doses of 4.5x10^5 PfSPZ or 9.0x10^5 PfSPZ to healthy Tanzanian children 1 to 5 years of age and infants 6 to 11 months of age, in each case compared to NS controls, will be evaluated. In addition, as an exploratory objective, controlled human malaria infection (CHMI) will be used to assess efficacy in adults three weeks following immunization.

Study Design: This is a single center trial with ten groups (Groups 1a/b: ages 18-45; Group 2a/b: ages 11-17; Group 3a/b: ages 6-10; Group 4a/b: ages 1-5; and Group 5b/c: ages 6months-11 months) each with 6 subjects receiving PfSPZ Vaccine and 3 subjects receiving NS and an eleventh smaller group (Group 5a: ages 6months-11months) with 3 subjects receiving PfSPZ Vaccine; two of these groups (Group 1a/b) contain adult volunteers and will have infectivity controls (CHMI 1 and 2) each having 3 subjects, after the vaccination phase of the study. The adult volunteers will undergo CHMI 3 weeks after the last immunization.

For the first immunization, two volunteers (out of six) in Group 1a will receive 9x10^5 of PfSPZ Vaccine by DVI as sentinels, to demonstrate safety and tolerability. At the same time, one (out of three) corresponding control volunteers will receive NS, in order to maintain blinding. Approximately 24 hours later, provided criteria for calling an ad hoc SMC meeting are not met, the remaining four volunteers in Group 1a will also receive a 9x10^5 PfSPZ dose of the vaccine and the remaining two placebo recipients will receive NS.

After review of at least +14 days post vaccination safety data for Group 1a by the SMC, if there are no significant safety concerns, two volunteers (out of six) in Group 1b will receive 1.8x10^6 PfSPZ, and two volunteers (out of six) in each of the Groups 2a and 3a will receive 9x10^5 PfSPZ, of the PfSPZ Vaccine, to demonstrate safety and tolerability, and each of these sentinel groups will be joined by one corresponding NS control in order to maintain blinding. Approximately 24 hours later, provided criteria for calling an ad hoc SMC meeting are not met, the remaining four volunteers in Group 1b will receive 1.8x10^6 PfSPZ and the remaining four volunteers in each of Groups 2a and 3a will receive 9x10^5 PfSPZ of the PfSPZ Vaccine, and the remaining placebo recipients will receive NS.

After review of at least +14 days post vaccination safety data for Groups 1b, 2a and 3a by the SMC, if there are no significant safety concerns, two volunteers (out of six) in each of the Groups 2b and 3b will receive 1.8x10^6 PfSPZ, those in Group 4a will receive 4.5x10^5 PfSPZ and all 3 volunteers in Group 5a will receive 2.7x10^5 PfSPZ of PfSPZ Vaccine, to demonstrate safety and tolerability, and each of the sentinel groups (two volunteers from Groups 2b, 3b and 4a) will be joined by one NS control in order to maintain blinding. Approximately 24 hours later, provided criteria for calling an ad hoc SMC meeting are not met, the remaining four volunteers in Groups 2b, 3b and 4a will receive their appropriate dose of PfSPZ Vaccine (1.8x10^6 PfSPZ, 1.8x10^6 PfSPZ, and 4.5x10^5 PfSPZ, respectively), and the placebo recipients will receive NS.

Escalation from the small group of infants, (Group 5a, n=3) receiving a single dose of 2.7x10^5 PfSPZ, to the full group (Group 5b, n=6) receiving three doses of 4.5x10^5 PfSPZ, will proceed without SMC review if criteria for calling an ad hoc SMC meeting are not met. However, if the criteria are met, an ad hoc SMC meeting will be called to review the data, and dose escalation to 4.5x10^5 PfSPZ will be postponed until the recommendations of the SMC are available. The interval between the 2.7x10^5 PfSPZ small group and the 4.5x10^5 PfSPZ larger group will be a minimum of three days.

After review of at least +14 days post vaccination, safety data for Groups 2b, 3b, 4a, 5a and 5b by the SMC, if there are no significant safety concerns, two volunteers (out of six) in each of the Groups 4b and 5c will receive 9x10^5 PfSPZ, to demonstrate safety and tolerability. At the same time, one (out of three) corresponding control volunteers will receive NS, in order to maintain blinding. Approximately 24 hours later, provided criteria for calling an ad hoc SMC meeting are not met, the remaining four volunteers in Group 4b and 5c will receive 9x10^5 PfSPZ dose of the vaccine, and the placebo recipients will receive NS.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, based on clinical and laboratory findings
* From the age 6 months to 45 years
* Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2; or adolescents, children and infants with Z-score of the selected indicator ([weight-for-height], [(height and BMI) for age]) category within ±2SD as detailed in protocol
* Long term (at least one year) or permanent residence in the Bagamoyo town or nearby villages
* Agreement to release medical information and to inform the study doctor concerning contraindications for participation in the study
* Willingness to be attended to by a study clinician and take all necessary medications prescribed during study period
* Agreement to provide contact information of a third party household member or close friend to study team
* Availability through mobile phone 24 hours during the entire study period
* Agreement not to participate in another clinical trial during the study period
* Agreement not to donate blood during the study period
* Able and willing to complete the study visit schedule over the study follow up period, including the hospitalizations required for protocol compliance
* Willingness to undergo HIV, hepatitis B (HBV) and hepatitis C (HCV) tests
* Volunteer (subjects 18 years of age and older) and parent or guardian signing informed consent (for subjects <18 years of age) is able to demonstrate their understanding of the study by responding correctly to 10 out of 10 true/false statements (in a maximum of two attempts for those who failed to respond correctly to all true/false statements in the first attempt)
* Signed written informed consent, in accordance with local practice, provided by adult volunteers, parents or legal representatives and relevant assent for children participants as applicable
* Free from malaria parasitaemia by blood smear at enrolment
* Free from helminth infections at enrolment, or diagnosed with helminthes and treated appropriately to eliminate infestation
* Female volunteers aged 9 years and above must be non-pregnant (as demonstrated by a negative serum pregnancy test), and provide consent / assent of their willingness to take protocol-defined measures not to become pregnant during the study and safety follow-up period

Exclusion Criteria:

* Previous receipt of an investigational malaria vaccine or drug in the last 5 years
* Participation in any other clinical study involving investigational medicinal products within 30 days prior to the onset of the study or during the study period
* History of arrhythmias or prolonged QT-interval or other cardiac disease, or Clinically significant abnormalities in electrocardiogram (ECG) at screening
* Positive family history in a 1st or 2nd degree relative for cardiac disease at age <50 years old
* A history of psychiatric disease
* Suffering from any chronic illness including; diabetes mellitus, cancer or HIV/AIDS
* Any confirmed or suspected immunosuppressive or immune-deficient condition, including asplenia
* History of drug or alcohol abuse interfering with normal social function
* The use of chronic immunosuppressive drugs or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids are allowed) and during the study period
* Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis
* Positive HIV, hepatitis B virus or hepatitis C virus tests
* Volunteers who are suspected as having clinically active TB by history or physical examination with positive QuantiFERON-TB Gold Test In-Tube assay
* Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, blood, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers
* Any medical, social condition, or occupational reason that, in the judgment of the investigator, is a contraindication to protocol participation or impairs the volunteer's ability to give informed consent, increases the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 6 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Incidence and type of Adverse Events | Post first immunization uptil 56 days post-CHMI or 56 days post-3rd immunization
  Incidence and type of adverse events (including breakthrough infections), vital signs, clinical laboratory assessments, physical examination findings post first immunization onwards.
  1. Occurrence of solicited symptoms during a 7-day surveillance period after vaccination (day of vaccination (Vx) and +7 days post vaccination)
  2. Occurrence of unsolicited symptoms during a 28-day surveillance period after each vaccination.
  3. Occurrence of serious adverse events during the study period.
  4. Occurrence of Pf infection of vaccine type detected at any point after the first vaccination (retrospectively determined).

SECONDARY OUTCOMES:
Level of Antibodies against Pf proteins in volunteer sera | Post first immunization uptil 56 days post-CHMI or 56 days post-3rd immunization
  1. Antibody titres to pre-erythrocytic stage and erythrocytic stage antigens[PfCSP, PfLSA-1, PfEBA-175 , PfMSP-1, PfMSP-5, EXP-1] by ELISA
  2. Antibody titres to Pf sporozoites, asexual and sexual erythrocytic stage parasites by IFA.
  3. Analysis of antibodies to proteins in the Pf proteome array chip.
Inhibitory Capacity of Volunteer Sera against in vitro Sporozoite Invasion of Hepatocytes | Post first immunization uptil 56 days post-CHMI or 56 days post-3rd immunization
  Capacity of sera from immunized volunteers to inhibit sporozoite invasion (ISI) of hepatocytes in vitro by ISI assay
Quantitation of cellular immune responses against Pf proteins in volunteers | Post first immunization uptil 56 days post-CHMI or 56 days post-3rd immunization
  1. Identification of number of vaccine induced PBMCs following Intracellular cytokine staining by flow cytometry after stimulation with PfSPZ or Pf-infected erythrocytes, peptide pools and P. falciparum infected primary human hepatocyte cell lines.
  2. Identification of numbers of vaccine induced CD4 and CD8 T cells following FluoroSpot assay after stimulation with PfSPZ or Pf-infected erythrocytes.
Whole genome expression profiles of volunteer | Post first immunization uptil 56 days post-CHMI or 56 days post-3rd immunization
  Human gene expression profiling focusing on immune response genes in volunteers

OTHER OUTCOMES:
Number of adult volunteers protected against CHMI following immunization | 28 days post CHMI
  Evidence of vaccine-mediated protection against CHMI 3 weeks after last immunization in Groups 1 (adults) by preventing blood stage infection for 28 days (as detected by blood smear analysis and qPCR) following CHMI.
Genetic profiles of Pf parasites | Screening uptil 56 days post-CHMI or 56 days post-3rd immunization
  Whole genome sequencing of Plasmodium falciparum following break through infections.

CONTACTS AND LOCATIONS:
Overall Officials: Said Jongo, MD, MMED, Principal Investigator — Ifakara Health Institute (IHI), Bagamoyo, Tanzania
Locations (1):
- Bagamoyo Research and Training center of the Ifakara Health Institute, Bagamoyo, Tanzania

REFERENCES:
- [Derived] Jongo SA, Church LWP, Mtoro AT, Schindler T, Chakravarty S, Ruben AJ, Swanson PA, Kassim KR, Mpina M, Tumbo AM, Milando FA, Qassim M, Juma OA, Bakari BM, Simon B, James ER, Abebe Y, Kc N, Saverino E, Fink M, Cosi G, Gondwe L, Studer F, Styers D, Seder RA, Schindler T, Billingsley PF, Daubenberger C, Sim BKL, Tanner M, Richie TL, Abdulla S, Hoffman SL. Increase of Dose Associated With Decrease in Protection Against Controlled Human Malaria Infection by PfSPZ Vaccine in Tanzanian Adults. Clin Infect Dis. 2020 Dec 31;71(11):2849-2857. doi: 10.1093/cid/ciz1152. PMID 31782768
- [Derived] Schindler T, Jongo S, Studer F, Mpina M, Mwangoka G, Mswata S, Ramadhani K, Sax J, Church LWP, Richie TL, Tanner M, Hoffman SL, Abdulla S, Daubenberger C. Two cases of long-lasting, sub-microscopic Plasmodium malariae infections in adults from coastal Tanzania. Malar J. 2019 Apr 29;18(1):149. doi: 10.1186/s12936-019-2787-x. PMID 31036014